CLINICAL TRIAL: NCT00594893
Title: A Prospective Randomized Trial of Mini Incision and 2-Incision Total Hip Arthroplasty
Brief Title: Study Comparing Mini-Incision Versus 2-Incision Approach for Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Craig J Delle Valle, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDV-05061503
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Hip; Arthroplasty; Minimally Invasive
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mini Incision Approach
  Interventions: Procedure: Mini Incision Approach
- 2 (Active Comparator): 2 Incision Approach
  Interventions: Procedure: 2 Incision Approach

INTERVENTIONS:
Procedure: Mini Incision Approach — Mini Incision Approach
  Arms: 1
Procedure: 2 Incision Approach — 2 Incision Approach
  Arms: 2

SUMMARY:
The purpose of the research is to determine if there is a difference between two of the commonly used less invasive techniques (surgical methods that use a smaller incision or cut in the skin) used to perform total hip arthroplasty (replacement of your painful hip with a new ball and socket). It is unclear which of these techniques is associated with a faster recovery and lower risk of complications.

DETAILED DESCRIPTION:
Recently, surgical techniques and surgical instruments have been developed to limit the dissection required to perform a total hip arthroplasty. Proponents of these procedures feel that it is associated with less perioperative blood loss, less pain and an accelerated recovery while critics have raised concerns that the more limited exposure may negatively impact component position and increase the risk of perioperative complications. Among less invasive surgical techniques, two of the different approaches utilized include a "mini-incision" posterior approach which aims to limit the amount of dissection associated with a standard posterior approach to the hip and a 2-incision technique which seeks to further limit soft tissue disruption by taking advantage of intermuscular planes and the use of fluoroscopic guidance.

While the mini-posterior approach utilizes an abbreviated exposure which is familiar to most surgeons, the 2-incision approach is a more novel approach and critics of this approach feel that its technically demanding nature may be associated with a higher risk of complications and component malposition. Proponents of the 2-incision approach feel that this approach is less invasive, more muscle sparing and leads to substantial improvements in patient rehabilitation and recovery with potential longer-term benefits in terms of improved function. The goal of this project is to compare the use of a mini-incision posterior approach and the 2-incision approach in primary total hip arthroplasty via a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hip osteoarthritis
* age greater than 18 years
* willingness to undergo a neuraxial anesthetic for the procedure
* female patient greater than one year postmenopausal, surgically sterile or using an accepted form of contraception

Exclusion Criteria:

* use of any medication that may impact platelet aggregation within 10 days of surgery
* chronic use of coumadin for anticoagulation
* the use of low molecular weight heparin postoperatively
* clinically significant systemic disease or laboratory abnormalities
* a primary hematologic disorder
* recent gastrointestinal or intracranial bleeding
* any contraindication to anticoagulant use
* history of previous ipsilateral hip surgery
* a body mass index of greater than 30
* significant hip deformity that precludes the use of standard implants
* use of ONLY general anesthetic during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain scores | Daily for 6 weeks postoperatively

SECONDARY OUTCOMES:
Functional milestones | daily for 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Craig J DellaValle, MD, Principal Investigator — Rush University Medical Center, Department of Orthopaedics
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Della Valle CJ, Dittle E, Moric M, Sporer SM, Buvanendran A. A prospective randomized trial of mini-incision posterior and two-incision total hip arthroplasty. Clin Orthop Relat Res. 2010 Dec;468(12):3348-54. doi: 10.1007/s11999-010-1491-5. Epub 2010 Jul 29. PMID 20668969